CLINICAL TRIAL: NCT01731912
Title: Degarelix Acetate Prior to Radiation Therapy
Brief Title: Degarelix Acetate Before and During Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bruce Montgomery, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7846; NCI-2012-02136 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD2; 7846 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2018-12

CONDITIONS: Prostate Adenocarcinoma; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (degarelix acetate, EBRT) (Experimental): Patients receive degarelix acetate SC on day 1. Treatment repeats every 4 weeks for up to 6 courses. Beginning at week 15, patients also undergo standard EBRT for 8.5 weeks.
  Interventions: Drug: Degarelix; Radiation: External Beam Radiation Therapy; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Degarelix — Given SC
  Other Names: FE200486; Firmagon
Radiation: External Beam Radiation Therapy — Undergo standard EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies how well degarelix acetate before and during radiation therapy works in treating patients with prostate cancer. Androgens can cause the growth of prostate cancer cells. Drugs, such as degarelix acetate, may lessen the amount of androgens made by the body. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving degarelix acetate together with radiation therapy may work better in treating prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of neoadjuvant degarelix (degarelix acetate) on prostate dihydrotestosterone (DHT) and testosterone levels.

SECONDARY OBJECTIVES:

I. To determine the effect of degarelix acetate on androgen-regulated gene expression and apoptosis as assessed by immunohistochemistry, complementary deoxyribonucleic acid (cDNA) microarray analysis and reverse transcriptase (RT)-polymerase chain reaction (PCR).

II. To determine the effect of degarelix acetate on follicle stimulating hormone (FSH) and FSH receptor expression in prostate cancer and surrounding microenvironment.

OUTLINE:

Patients receive degarelix acetate subcutaneously (SC) on day 1. Treatment repeats every 4 weeks for up to 6 courses. Beginning at week 15, patients also undergo standard external beam radiation therapy (EBRT) for 8.5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Written authorization for use and release of health and research study information has been obtained
* Histologically proven adenocarcinoma of the prostate
* Patients must be candidates for short or long term androgen deprivation in combination with external beam radiation therapy (RT) based on the following criteria:

  * Intermediate risk disease: T2b/c, or Gleason 7, or prostate-specific antigen (PSA) 10-20
  * High risk disease: Gleason 8-10, or PSA > 20, or T3/4
* Patients may not have received any prior pharmacologic therapy or RT for prostate cancer
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the androgen axis will be determined following review of their case by the principal investigator
* Patients must allow biopsy at the time of fiducial placement

Exclusion Criteria:

* Patients may not be receiving any investigational agents
* Patients who are currently receiving active therapy for other neoplastic disorders will not be eligible
* Patients with histologic evidence of small cell carcinoma of the prostate will not be eligible
* Patients with hypogonadism or severe androgen deficiency as defined by serum testosterone less than 100 ng/dL will not be eligible
* History of pituitary dysfunction
* Patients who are receiving any androgens, estrogens or progestational agents, or who received any of these agents within the 6 months prior to evaluation will not be eligible
* Patients who are taking drugs which affect androgen metabolism (e.g. spironolactone, ketoconazole, finasteride, dutasteride) will not be eligible; patients who received any of these agents within the 6 months prior to evaluation will be reviewed for eligibility by the principal investigator on a case by case basis
* Patients with inflammatory bowel disease or other autoimmune conditions which might affect the radiated colon or rectum
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia which is symptomatic or requires active therapy, recent deep venous thrombosis, pulmonary emboli, cerebrovascular accident or ischemia will not be eligible
* Patients with dementia/psychiatric illness/social situations that would limit compliance with study requirements or would prohibit the understanding and/or giving of informed consent will not be eligible
* Patients with medical conditions, which, in the opinion of the investigators, would jeopardize either the patient or the integrity of the data obtained will not be eligible
* Other active malignancy, except non-melanoma skin cancer and superficial bladder cancer
* Patients unwilling to use contraceptives while on study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montgomery, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 started therapy. 14 completed therapy
Groups:
- Degarelix: Patients receive 3 months of degarelix prior to radiation and then for 3 months during radiation. Subsequent therapy is determined by the treating physician
Period: Overall Study
Arm/Group | Degarelix
Started | 16
Completed | 14
Not Completed | 2
Not completed — noncompliance | 2

BASELINE CHARACTERISTICS:
Arm/Group | Degarelix
Number analyzed (Participants) | 16
Age, Continuous [Median (Standard Deviation); unit: years] | 65 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Tissue Levels of DHT in Prostate Tissue as Measured by Mass Spectometry
Description: Differences in tissue androgen levels between this group and historical comparisons will be evaluated by performing a one-way analysis of variance (ANOVA), followed by pair-wise two-sample t-tests to determine which groups are statistically different.
Time Frame: At week 24
Population: Tissue DHT at 24 weeks
Measure: Median (Standard Deviation); unit: pg/mg
Arm/Group | Degarelix
Number analyzed (Participants) | 14
pg/mg | 0.6 (0.34)

2. Primary Outcome: Tissue Levels of Testosterone in Prostate Tissue as Measured by Mass Spectometry
Time Frame: At week 24
Population: Tissue testosterone levels at 24 weeks
Measure: Median (Standard Deviation); unit: pg/mg
Arm/Group | Degarelix
Number analyzed (Participants) | 14
pg/mg | 0.17 (0.13)

ADVERSE EVENTS:
Description: Degarelix is FDA approved for hormonal treatment of prostate cancer and concurrent administration with radiotherapy in this study and is not considered outside of the standard of care; reporting adverse events was not required. Per the protocol AE reporting was not planned, therefore no AE data was collected.
Arm/Group | Degarelix
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes